CLINICAL TRIAL: NCT05506306
Title: Multitissular Effect of Vertical Mobilization Using the Exoskeleton AtalanteTM in Neurological Chair- or Bed-bound Patients
Acronym: VERTEXO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Henri Mondor University Hospital (Other)
Responsible Party: Principal Investigator, ETIENNE SAVARD, hospital practicioner, Henri Mondor University Hospital
Other Study IDs: 2022-A0134142
Record Dates: First submitted 2022-08-08; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Neurologic Disorder
MeSH Terms: conditions — Nervous System Diseases | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment — Clinical, biological and imagery before and after 6 weeks of using AtalanteTM exoskeleton

SUMMARY:
Background and aim: Sustained bed rest impairs many bodily functions. Verticalization restores gravitational challenge and the use of several organs. The Atalante™ exoskeleton (Wandercraft) is the only self-balanced exoskeleton, which allows walking without canes. We assessed multi-tissular effects of mobile reverticalization using Atalante™ in neurological bed- or wheelchair-bound patients.

Methods: Observational cohort study. Inclusion criteria: bed- or wheelchair-bound for >2 weeks and <1 hour per day of stance, due to a central neurological disorder. Sessions with exoskeleton were 3/week, integrated in routine care. Data collected at baseline and after eight weeks (W8) included: cardiovascular (echocardiography, EKG, blood pressure lying and standing), pulmonary (spirometry), bone (densitometry, biochemical markers), bowels (daily stool frequency, Bristol Stool Scale), urinary (urinary flow, postmictional residual volume, urinary symptom profile questionnaire, USP), cognitive (trail making test, TMT-B), anxiety and depression (HAD), and quality of life (SF12).

Results will be presented at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* inpatient in neurorehabilitation
* neuroligical lesion
* chair or bed bound more than 23h/24h and more than 2 weeks
* over 18 years old

Exclusion Criteria:

* spasticity over 3 on MAS
* any porotic fracture
* heel pressure sore
* Height > 150 cms, > 190 cms
* Weight < 30 kgs > 90 kgs
* recent thoracic or abdominal surgery
* pregnancy
* range of motion aloud to use the exoskeleton

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients Neurological patients non-walking
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Mean Hospital Anxiety and Depression scale at 6 weeks | baseline and 6 weeks
  HAD
Change from Baseline in the Mean Sonographic Cardiac index at 6 weeks | baseline and 6 weeks
Change from Baseline in the Mean first second of forced expiration at 6 weeks | baseline and 6 weeks
  FEV1
Change from Baseline in the Mean serum sclerostin at 6 weeks | D0 and D45
Change from Baseline in the Mean stool frequency at 6 weeks | baseline and 6 weeks
Change from Baseline in the Mean maximal urine flow rate at 6 weeks | D0 and D45
Change from Baseline in the Mean Trail Making Test B at 6 weeks | baseline and 6 weeks
  TMT-B

SECONDARY OUTCOMES:
Change from Baseline in the Mean blood pressure at rest at 6 weeks | baseline and 6 weeks
Change from Baseline in the Mean stroke volume at 6 weeks | baseline and 6 weeks
  assessed by sonography
Change from Baseline in the Mean filling pressure at 6 weeks | baseline and 6 weeks
  assessed by sonography
Change from Baseline in the Mean Forced vital capacity at 6 weeks | baseline and 6 weeks
  FVD is assessed by spirometry
Change from Baseline in the Mean serum calcium at 6 weeks | baseline and 6 weeks
Change from Baseline in the Mean serum creatine phosphokinase at 6 weeks | baseline and 6 weeks
  CPK
Change from Baseline in the Mean serum parathormone at 6 weeks | baseline and 6 weeks
  PTH
Change from Baseline in the Mean serum D vitamin at 6 weeks | baseline and 6 weeks
Change from Baseline in the Mean serum phosphatases alcalines at 6 weeks | baseline and 6 weeks
  PAL
Change from Baseline in the Mean serum carboxy-terminal collagen crosslinks at 6 weeks | baseline and 6 weeks
  CTX
Change from Baseline in the Mean serum Tartrate-resistant acid phosphatase 5b at 6 weeks | baseline and 6 weeks
  TRAP5b
Change from Baseline in the Mean serum osteocalcin at 6 weeks | baseline and 6 weeks
Change from Baseline in the Mean urin calcium at 6 weeks | baseline and 6 weeks
  bone densitometry
Change from Baseline in the Mean bone densitometry at 6 weeks | baseline and 6 weeks
Change from Baseline in the Mean bristol stool scale at 6 weeks | baseline and 6 weeks
Change from Baseline in the Mean voided volume at 6 weeks | baseline and 6 weeks
Change from Baseline in the Mean post void residue at 6 weeks | baseline and 6 weeks
Change from Baseline in the Mean urinary symptom profile SCORE at 6 weeks | baseline and 6 weeks
  USP
Change from Baseline in the Mean fatigue severity SCALE at 6 weeks | baseline and 6 weeks
  FSS
Change from Baseline in the Mean trail making test A at 6 weeks | baseline and 6 weeks
  cognitive assessment
Change from Baseline in the Mean fluence at 6 weeks | baseline and 6 weeks
  cognitive assessment
Change from Baseline in the Mean span at 6 weeks | baseline and 6 weeks
  cognitive assessment
Change from Baseline in the Mean Medical Outcome Study Short Form 12 at 6 weeks | baseline and 6 weeks
  quality of life assessment

IPD SHARING:
Plan to Share IPD: Undecided